CLINICAL TRIAL: NCT06815185
Title: Rehabilitation Counselling for Patients with Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ReF2202
Record Dates: First submitted 2025-01-22; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-09

CONDITIONS: Fibrosis, Pulmonary
Keywords: rehabilitation counselling
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a rare chronic progressive disease of unknown etiology that affects physical and emotional well-being. It is characterized by irreversible loss of lung function due to fibrosis, which manifests itself with cough, dyspnea, and impaired quality of life. Lung transplantation is limited to a minority of patients and patients receive anti-fibrotic therapy in addition to supportive/palliative treatments. In light of the broad definition of pulmonary rehabilitation, and by virtue of the multidisciplinary nature of the process, the present study aims to observe the effects of the rehabilitation counseling offered to patients who attend the IPF clinic at the Pneumology Operating Unit of the IRCCS Company Bologna University Hospital, as part of the Intercompany PDTA (diagnostic therapeutic care path) for Pulmonary Fibrosis: the Intercompany PDTA for patients suffering from idiopathic pulmonary fibrosis involves a multidisciplinary approach which, also through therapeutic education/counselling, aims among others to "Offer the patient the opportunity to participate in clinical studies to increase knowledge about the disease and/or have access to innovative treatments". Primary objectives

1. Evaluate the effectiveness of the rehabilitation intervention contained in the PDTAI (Intercompany diagnostic therapeutic care path )
2. Evaluate the improvement in functional capacity and cardiorespiratory endurance.

   Secondary objectives
3. Evaluate the progress and evolution of the pathology.
4. Evaluate the emotional burden of the caregiver in caring for the individual suffering from IPF
5. Evaluate the improvement in quality of life.
6. Evaluate the change in disability.
7. Evaluate the patient's fatigue and its evolution over the course of the disease. Fatigue is associated with dyspnea, impacts daily living activities and quality of life.
8. Evaluate the progress and evolution of dyspnea at rest and in relation to the performance of common daily activities.

The study plans to enroll 40 patients newly diagnosed with IPF

Inclusion criteria:

* adulthood ≥18 years
* Obtaining the patient's informed consent

Exclusion criteria:

* diagnosis of cancer in the active phase
* Situations of clinical instability, of clinical worsening such as to deem the individual unsuitable for treatment because they are no longer able to go to follow up visits The included patients will receive the therapeutic education brochure from the physiotherapist and will be trained to perform the exercises during hospital visits. The physiotherapist will be able to evaluate and modify the retraining program based on the user's response according to the principles based on the individualized rehabilitation project. The direct comparison with the user allows to obtain a functional improvement adapted to the needs and performance of the person but at the same time, according to the principles of empowerment, helps the subject to become aware of their functional limits and address them with a more personalized.

The sessions will be planned following the criteria of frequency, intensity, time and type of exercise:

Frequency: one meeting/every fifteen days in the first month and one meeting every fifteen days (+/- five days) in the second and third months.

Intensity: sixty minutes (with mBorg three dyspnea and minimum peripheral saturation 88%) Time: sixty minutes Type of treatment: exercises from the therapeutic education brochure.

Endpoints measures:

1. % of patients participating in the physiotherapy session programme. It is expected that at least 80% of the total enrolled participants will participate in the proposed session cycle.
2. Six Minute Walking Test. This test is validated for multiple pathologies, including idiopathic pulmonary fibrosis.
3. % Survival of IPF patients.
4. Caregiver Strain Index.
5. EuroQoL scale.
6. Barthel Index Dyspnea.
7. Fatigue Assessment Scale.
8. Modified British Medical Research Council.

ELIGIBILITY:
Inclusion Criteria:

* age>/= 18 years old;
* Obtaining the patient's informed consent

Exclusion Criteria:

* Diagnosis of active cancer
* Situations of clinical instability, clinical aggravation such as to consider unsuitable the individual to treatment because he or she is no longer able to go to follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients newly diagnosed with IPF will be enlisted but only who comply with the criteria for rehabilitation care:
  6MWT -meters ≥ 200 (Functionalcapacity); O2 therapy (Lt/min.) ≤ 3; Resting SpO2 ≥ 91% (Peripheraloxygensaturation); FVC (% predicted) ≥ 50% (Pulmonaryfunction); DLCO ≥ 30%(Pulmonaryfunction); mBorg at rest (score) ≤ 4 (Dyspnea); mMRC (score) ≤ 3 (Dyspnea)
  As IPF is a rare disease, it is estimated that 20 patients/year can be enrolled on the basis of of the cases relating to previous years, therefore, considering the two years of enrolment, we expect to be able to enroll a total number of 40 patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the rehabilitation intervention contained in the PDTAI (Inter-company diagnostic and therapeutic pathway) | 56 months
  % of patients participating in the physiotherapy session program, at least that 80% of the total enlisted participate in the cycle of sessions proposed.
Improvement of functional capacity and cardiorespiratory endurance | 56 months
  Six Minute Walking Test (6MWT). This test is validated for multiple pathologies, including idiopathic pulmonary fibrosis. MCID range from 21.7 to 45 meters. One reduction of more than 50 meters in 6 months increases mortality by three times

SECONDARY OUTCOMES:
% Survival of patients with IPF. | 56 months
  % Survival of patients with IPF.
Caregiver Strain Index | 56 months
  Evaluate the emotional burden of the caregiver in assisting the affected person by IPF
EuroQoL scale (EQ-5D-5L) | 56 months
  Evaluate the improvement in quality of life
Barthel Index Dyspnea | 56 months
  Evaluate the modification of disability
Fatigue Assessment Scale (FAS) | 56 months
  Evaluate the patient's fatigue and its evolution during the course of the disease. Fatigue is associated with dyspnea, impacts daily life activities and quality of life.
Modified British Medical Research Council (mMRC) | 56 months
  Evaluate the trend and evolution of dyspnea at rest and in relation to completion of common daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Enrica Cavalli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No